CLINICAL TRIAL: NCT04804657
Title: Effects of Sage Extracts on Cognitive Function During Aerobic Exercise in Healthy Individuals
Brief Title: Effects of Sage Extracts on Cognitive Function During Aerobic Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Burgundy (Other)
Responsible Party: Principal Investigator, Nicolas Babault, Principal investigator, University of Burgundy
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: CEP2101
Record Dates: First submitted 2021-01-26; First posted 2021-03-18 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Healthy
Keywords: cycling; cognition; sage; memory; fatigue
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sage extract (Active Comparator): Two hours before the endurance test, participants were asked to absorb two capsules of sage extracts (600mg each - cognivia™)
  Interventions: Dietary Supplement: Sage extracts Cognivia
- placebo (Placebo Comparator): Two hours before the endurance test, participants were asked to absorb two capsules of placebo (similar appearance than active comparator).
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Sage extracts Cognivia — Cognivia is composed of 400 mg of aqueous extract from Salvia officinalis and the remaining 200 mg contained 50 µL of Salvia lavandulaefolia essential oil and encapsulated with gum acacia. It will be administrated the the morning before the endurance test (oral administration).
  Arms: Sage extract
Dietary Supplement: Placebo — Made with maltodextrin. It will be administrated the the morning before the endurance test (oral administration).
  Arms: placebo

SUMMARY:
Extracts of sage have been reported to interact with central nervous system (CNS) mechanisms relevant to cognitive performance but, to date, no trial has clearly demonstrated the possible effects in healthy individuals in fatiguing conditions. The current study investigates the effects of this supplementation in healthy males and females versus placebo on cognition, heart rate and perceived exertion, during a fatiguing cycling exercise.

DETAILED DESCRIPTION:
Healthy males and females will be tested in fresh and fatiguing conditions to mimic individuals at the beginning or during a competition where cognitive function are important for decision making for example. Tests will be conducted during the warm-up (fresh), during fatiguing situations (during two consecutive 10-minutes pedaling exercises) and during recovery. Tests will include a reverse digit memory test (from 3 to 7 digits), a stroop test, a simple reaction time test. Moreover, heart rate and rating of perceived exertion will be quantified.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index lower than 27 and waist size lower than 94 cm
* physical activity higher than 3 hours a week
* written informed consent

Exclusion Criteria:

* more than 12 hours training a week
* asthmatic, smokers or under medicinal drugs
* dietary supplement, sports drink, special dietary food or functional food, of any kind, liable or presented as liable to enhance physical performances

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-03-15 (Actual)

PRIMARY OUTCOMES:
Memory | During the 10-minutes warm-up, immediately after the first 10-minutes fatiguing exercise, after the second 10-minutes fatiguing exercise and after a five minutes recovery period
  Changes in percent number of correct answers during a reverse digit immediate memory test

SECONDARY OUTCOMES:
Heart rate | At rest, at the end of the 10-minutes warm-up, at the end of the first 10-minutes fatiguing exercise, at the end of the second 10-minutes fatiguing exercise, after 5 minutes of recovery
  Changes in heart rate using a polar belt (in beats per minutes)
Rating of perceived exertion | At rest, at the end of the 10-minutes warm-up, at the end of the first 10-minutes fatiguing exercise, at the end of the second 10-minutes fatiguing exercise, after 5 minutes of recovery
  Changes in rating of perceived exertion using a visual analogic scale (1-10)
Reaction time | During the 10-minutes warm-up, immediately after the first 10-minutes fatiguing exercise, after the second 10-minutes fatiguing exercise and after a five minutes recovery period
  Changes in reaction time between a visual signal and manual action
Stroop performance | During the 10-minutes warm-up, immediately after the first 10-minutes fatiguing exercise, after the second 10-minutes fatiguing exercise and after a five minutes recovery period
  Changes in percent number of correct answers during a stroop test
Stroop reaction time | During the 10-minutes warm-up, immediately after the first 10-minutes fatiguing exercise, after the second 10-minutes fatiguing exercise and after a five minutes recovery period
  Changes in reaction time during the stroop test

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Babault, PhD, Principal Investigator — University of Burgundy
Locations (1):
- Centre d'Expertise de la Performance, Dijon, France

IPD SHARING:
Plan to Share IPD: No